CLINICAL TRIAL: NCT03922061
Title: Phase I Evaluation of the Safety, Reactogenicity and Immunogenicity of Fractional-dose Inactivated Polio Vaccine (fIPV) Given Intradermally With Double Mutant [LT(R192G/L211A)] Enterotoxigenic Escherichia Coli Heat Labile Toxin (dmLT) Adjuvant
Brief Title: Evaluation of Safety, Reactogenicity and Immunogenicity of Fractional-dose Inactivated Polio Vaccine (fIPV) Given Intradermally With Double Mutant Enterotoxigenic Escherichia Coli Heat Labile Toxin (dmLT) Adjuvant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Kelly Cowan, Assistant Professor of Pediatrics, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHRMS 19-0048
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Polio
Keywords: inactivated polio vaccine (IPV); fractional-dose inactivated polio vaccine (fIPV); double mutant [LT(R192G/L211A)] Enterotoxigenic E coli heat toxin (dmLT)
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- fIPV-dmLT (Experimental): fractional-dose inactivated polio vaccine (fIPV) given intradermally with double mutant [LT(R192G/L211A)] Enterotoxigenic Escherichia coli heat labile toxin (dmLT) adjuvant
  Interventions: Biological: dmLT; Biological: fIPV
- fIPV (Active Comparator): fractional-dose inactivated polio vaccine (fIPV) given intradermally
  Interventions: Biological: fIPV

INTERVENTIONS:
Biological: dmLT — double mutant [LT(R192G/L211A)] Enterotoxigenic Escherichia coli heat labile toxin (dmLT)
  Arms: fIPV-dmLT
Biological: fIPV — fractional-dose inactived polio vaccine

SUMMARY:
Polio is a serious disease that can cause paralysis and death. It is caused by a virus and can be prevented by vaccine. The World Health Organization's (WHO) Global Polio Eradication Initiative is trying to get rid of all polio disease around the world. Researchers want to help by testing a new vaccine.

In many countries, people are vaccinated with oral polio vaccine (OPV) given by mouth during childhood. OPV is good at giving immunity (protection from polio) in the body and the gastrointestinal (GI) tract. Immunity in the GI tract is called mucosal immunity. The downsides of using OPV are that it can be shed into the environment in people's feces after vaccination where it can infect people who are not vaccinated, and it can cause paralysis in 2-4 of every one million children vaccinated with OPV. The United States (U.S.) stopped giving any OPV to people for vaccinations in the 1990's. Since then, a polio vaccine called inactivated polio vaccine (IPV) is given as an injection for routine childhood immunizations in the U.S. You cannot get polio infection from IPV and it will not be shed into the environment.

In 2016, the WHO started a plan to help other countries gradually get rid of OPV. The downside of using IPV by itself is that, unlike OPV, it doesn't give enough mucosal immunity to protect people living in places where there is still polio. There are also supply shortages of IPV, which is a problem if there are outbreaks of polio. For the supply of IPV to help more people, it is safe and effective to use a tiny dose of IPV injected under the top layer of skin (intradermal or ID injection) rather than getting the full dose in the muscle. This is called a fractional dose of IPV, or fIPV.

To help stop using OPV globally, a better fIPV vaccine is needed. fIPV vaccine needs a substance to help stimulate a mucosal immune response. dmLT is a substance that has been shown to stimulate a mucosal immune response. It has been shown to be safe and effective in both humans and animals, both by itself and when given with other vaccines.

This study will test a mixture of fIPV-dmLT given intradermally (under the outer layer of the skin). This is the first study done in humans to give this combination intradermally. The IPV vaccine has already been approved by the FDA. The fIPV-dmLT vaccine has not been approved by the FDA.

DETAILED DESCRIPTION:
This single site study conducted at The University of Vermont will enroll 30 healthy male and female adult volunteers aged 18-45 years with no history of oral polio vaccination for a Phase I randomized controlled double-blind trial evaluating the safety, reactogenicity and immunogenicity of a single dose of fIPV-dMLT versus a single dose of fIPV administered intradermally. Study volunteers will be screened with eligible volunteers enrolled who will randomized to receive a single dose of fIPV-dmLT or fIPV (2:1) on study day 0. The primary study objective is to determine the safety and reactogenicity of a single dose of adjuvanted fIPV-dmLT vaccine in healthy adults, as assessed by the frequency of systemic and local injection site adverse reactions (ARs) defined as vaccine-related adverse events (AEs), graded by severity, occurring within 28 days of dosing. Secondary objectives are to determine the safety of a single dose of adjuvanted fIPV-dmLT vaccine in healthy adults, as assessed by the percentage of subjects with at least one vaccine-related serious adverse event (SAE) occurring within 28 days of dosing. In addition, the systemic immune response to a single dose of vaccine in healthy adults, as assessed by poliovirus-specific serum neutralizing antibody responses in fIPV-dmLT recipients versus fIPV only recipients will be examined.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female age 18-45 years, inclusive
2. Signed informed consent form prior to initiation of any study activity
3. Good general health as determined by review of medical history and physical exam
4. Agrees to complete all study visits and procedures for the duration of the study
5. Receipt of childhood vaccine series of Inactivated Polio Vaccine with verification of immunization record. American College of Immunization Practices (AICP) required that OPV use be discontinued by January 2000. Therefore, polio vaccines given after January 2000 in the U.S. are known to be IPV. If the documentation is unclear of the type of polio vaccine given between 1998 and 2000, additional confirmation of the type should be attempted to determine eligibility.
6. Agrees to storage of specimens for future research
7. Females of child bearing potential only: willing to use effective contraception from the following reliable methods through the first 28 days of the study: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, and intrauterine device. All female subjects will be considered as having childbearing potential except for those who have had a hysterectomy or tubal ligation or have no internal female organs. Transgender men who have internal female organs will be considered of childbearing potential and should be willing to use effective contraception during the trial. Exception: females who have sex with females (exclusively) and have no intention of conceiving a child during the study will not be required to use contraception.

Exclusion Criteria:

1. History of receipt of any oral polio vaccine. Subjects will be required to present their childhood immunization record during the screening process. Subjects will be excluded if the immunization record indicates receipt of any dose of oral polio vaccine or if only 'polio vaccine' is listed on the record without specifying whether oral or inactivated polio vaccine was administered.
2. Currently lactating, breastfeeding or pregnant.
3. Clinical laboratory values ≥ Grade 2 on hematology or comprehensive metabolic panel, as defined in this protocol.
4. Febrile illness (≥38.0°C (100.4°F) or acute gastroenteritis within 48 hours prior to administration of IP
5. History of antimicrobial treatment in the 2 weeks before administration of IP
6. Receipt of a live vaccine within 28 days or a killed vaccine within 14 days prior to inoculation, or anticipated receipt of any vaccine during the 28 days following inoculation.
7. History of a severe allergic reaction or anaphylaxis
8. History of Guillian-Barre Syndrome
9. Known history of hypersensitivity to any component of IPV to include: 2-phenoxyethanol, formaldehyde, neomycin, streptomycin, and polymyxin B
10. Self-reported or suspected immunodeficiency, or receipt of immunosuppressive therapy within the preceding 6 months, or long-term systemic corticosteroid therapy. An immunosuppressive dose of corticosteroids (excluding topical or nasal) is defined as >10 mg of prednisone equivalent per day for >14 days.
11. Asplenia
12. Receipt of blood products within the past 6 months, including transfusions or immunoglobulin, or anticipated receipt of any blood products or immunoglobulins during the 28 days following inoculation
13. Anticipated receipt of any investigational agent in the 28 days before or after receipt of investigational product
14. Abnormal routine bowel habits as defined by fewer than three stools per week in the past 6 months
15. Regular use (weekly or more often) of laxatives, anti-diarrheal, anti-constipation, or antacid therapy
16. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease based on history and physical exam. This includes any chronic medical condition (examples include diabetes mellitus, hypertension, autoimmune disorders, cardiovascular and renal diseases).
17. Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the subject's ability to understand and cooperative with the requirements of the study protocol.
18. Any other condition that, in the opinion of the study clinician, would jeopardize the safety or rights of a subject participating

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
frequency of systemic and local injection (safety and reactogenicity) | Events occuring within 28 days of dosing
  frequency of systemic and local injection site adverse reactions (ARs) defined as vaccine-related adverse events (AEs), graded by severity

SECONDARY OUTCOMES:
percentage of subjects with at least one serious adverse event (secondary-safety) | Events occuring within 28 days of dosing
  percentage of subjects with at least one serious adverse event (SAE) occurring within 28 days of dosing will be summarized with severity, relationship to vaccine, and outcome
Systemic immunogenicity | Any timepoint up to day 28 post-vaccination
  Proportion of participants showing at least a 4-fold boost in polio-specific serum neutralizing antibodies compared to baseline (Day 0) in fIPV-dmLT recipients vs. fIPV alone

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Cowan, M.D., Principal Investigator — University of Vermont; Beth Kirkpatrick, M.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crothers JW, Ross Colgate E, Cowan KJ, Dickson DM, Walsh M, Carmolli M, Wright PF, Norton EB, Kirkpatrick BD. Intradermal fractional-dose inactivated polio vaccine (fIPV) adjuvanted with double mutant Enterotoxigenic Escherichia coli heat labile toxin (dmLT) is well-tolerated and augments a systemic immune response to all three poliovirus serotypes in a randomized placebo-controlled trial. Vaccine. 2022 Apr 26;40(19):2705-2713. doi: 10.1016/j.vaccine.2022.03.056. Epub 2022 Mar 30. PMID 35367069

DOCUMENTS (1):
  • Informed Consent Form (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT03922061/ICF_000.pdf